CLINICAL TRIAL: NCT03591913
Title: Comparison Between Preoperative and Postoperative Sublingual Misoprostol for Prevention of Postpartum Blood Loss in Cesarean Section : a Randomized Clinical Trial
Brief Title: Preoperative and Postoperative Sublingual Misoprostol for Prevention of Postpartum Blood Loss in Cesarean Section
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed Abbas, Principal investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: MISOCS
Record Dates: First submitted 2018-07-08; First posted 2018-07-19 (Actual); Last update posted 2018-09-18 (Actual); Status verified 2018-09

CONDITIONS: Postpartum Hemorrhage
MeSH Terms: conditions — Postpartum Hemorrhage | interventions — Misoprostol

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study group (Experimental): will receive sublingual misoprostol immediately after urinary catheterization and before skin incision
  Interventions: Drug: Misoprostol
- control group (Active Comparator): will receive sublingual misoprostol immediately after skin closure
  Interventions: Drug: Misoprostol

INTERVENTIONS:
Drug: Misoprostol — Oral tablets

SUMMARY:
Cesarean section is one of the most common major surgical operations among women. In 2015, the incidence of cesarean section in Woman Health Hospital in Assiut University accounts for 51.3 % of all deliveries

ELIGIBILITY:
Inclusion Criteria:

* All pregnant women who will undergo elective lower segment cesarean section
* term ( ≥ 37 weeks)
* normal fetal heart tracing.

Exclusion Criteria:

* Placenta previa-Rupture uterus
* Classical cesarean section
* Preterm delivery
* Hypertensive disorders of pregnancy
* Bleeding tendency
* Previous history of postpartum hemorrhage
* Concurrent anticoagulant therapy
* Concurrent long-term use of steroids
* Fetal distress
* Antepartum haemorrhage

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 500 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2018-08-01 (Actual); Study Completion 2018-09-01 (Actual)

PRIMARY OUTCOMES:
mean intraoperative blood loss | 24 hours
  Blood loss estimation will commence immediately following the skin incision

CONTACTS AND LOCATIONS:
Locations (1):
- Ahmed Abbas, Assiut, Cairo Governorate, Egypt